CLINICAL TRIAL: NCT03121807
Title: A Pilot Study of Home Parenteral Nutrition for Malnourished Patients With Unresectable Stage IV Gastric Receiving Salvage Chemotherapy
Brief Title: Home Parenteral Nutrition for Malnourished Unresectable Stage IV Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jaw-Yuan Wang, MD, PhD, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KMUHIRB-20130271
Record Dates: First submitted 2017-01-04; First posted 2017-04-20 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Gastric Cancer
Keywords: home parenteral nutrition
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home parenteral nutrition (Experimental): Home parenteral nutrition with 910 kcal/day , including 33 g amino acid/day, 120 g glucose/day, 30 g lipid/day and electrolyte, micro-element and vitamin according to the nutritional status of subjects and followed the standard procedure of the hospital (Oliclinomel N4 Per bag 1.5 L), was infused continuously daily in an infusion time ranged between 18-24 hours.
  Patients received 85 mg/m2 oxaliplatin and 200 mg/m2 leucovorin as a 2-h intravenous infusion on day 1, followed by 2400 mg/m2 5Fluorouracil as a 46-h continuous infusion. This regimen is repeated every 14 days as a cycle.
  Interventions: Other: Oliclinomel N4 Per bag 1.5 L; Drug: Oxaliplatin; Drug: 5Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Other: Oliclinomel N4 Per bag 1.5 L — Home parenteral nutrition with 910 kcal/day , including 33 g amino acid/day, 120 g glucose/day, 30 g lipid/day and electrolyte, micro-element and vitamin according to the nutritional status of subjects and followed the standard procedure of the hospital (Oliclinomel N4 Per bag 1.5 L), was infused continuously daily in an infusion time ranged between 18-24 hours.
Drug: Oxaliplatin
  Other Names: Eloxatin
Drug: 5Fluorouracil
  Other Names: 5Fu
Drug: Leucovorin
  Other Names: folinic acid

SUMMARY:
This survey is a single arm study to assess the effect of home parenteral nutrition on overall survival, cycles of salvage chemotherapy completed, side effects of salvage chemotherapy, quality of life, nutritional status, functional status, inflammatory status and complications of HPN in malnourished unresectable metastatic gastric cancer (mGC) patients in a single medical center. It is expected that about 20 subjects will be recruited during an estimated period of 48 months.

DETAILED DESCRIPTION:
Objectives:

1. Primary Objective:

   The primary end points are overall survival and cycles of salvage chemotherapy completed of malnourished patients in unresectable mGCs
2. Secondary Objectives:

Side effects of salvage chemotherapy, quality of life, nutritional status, performance status, inflammatory status, safety and complications of HPN. The visit time schedules are at the time of enrollment before HPN is delivered, and at the beginning of every cycle of salvage chemotherapy

Patient Selection and Enrollment:

Twenty patients are planed to be enrolled

Drop out The following reasons may consider to withdrawing a patient from the study

1. Intolerance adverse events
2. Patient will exceed defined safety cut-off values e.g. increase of a certain amount of a laboratory parameter.
3. Violation of study protocol
4. Withdraw of informed consent.

Study duration and dates The study of this protocol is expected to be approximately 24 months, with a subject recruitment period of 18 months (proposed to start in Sep 2014 and end in Sep 2018). The duration of the study or period of recruitment may vary.

Treatment duration HPN is administered till resolution of malnutrition or till patient dies

.

ELIGIBILITY:
Inclusion Criteria:

1. Histology confirmed adenocarcinoma of stomach.
2. Stage IV (AJCC 7.0)
3. Malnourished patients with nutritional risk index (NRI) < 97.5. NRI= 1.59 x serum albumin level (g/L) + 0.417 x (current weight/usual weight) x 100
4. Adequate organ function as defined by the following criteria:

   * absolute neutrophil count (ANC) > or =1500 cells/mm3;
   * platelets > or =60,000 cells/mm3
   * hemoglobin > or =8.0 g/dL
   * AST and ALT < or =3.0 x upper limit of normal (ULN), unless there are liver metastases in which case AST and ALT< or =5.0 x ULN;
   * total bilirubin < or =2.0x ULN
   * serum creatinine < or =2.0 x ULN or calculated creatinine clearance > or =60 mL/min
5. Male or female, age > or = 20 years and < 80 years.
6. Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment.
7. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.

Exclusion Criteria:

1. Known allergy to components of studied parenteral nutrition.
2. Acute shock or collapse.
3. Known diabetic ketoacidosis 7 days prior to randomization.
4. Unstable conditions (e.g. uncompensated diabetes mellitus, acute myocardial infarction, embolism, metabolic acidosis, severe sepsis and hypotonic dehydration).
5. General contraindications to infusion therapy: acute pulmonary edema, hyperhydration, uncompensated cardiac insufficiency.
6. Investigator judges as subjects to be inappropriate for the clinical study (e.g., patient with severe complications)
7. Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
8. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness.
9. Participation in another clinical study with an investigational drug or an investigational medical device within 1 month prior to start of the study or during the study.
10. Female patients who are pregnant or lactating, or men and women of reproductive potential not willing or not able to employ an effective method of birth control/contraception to prevent pregnancy during treatment and for 6 months after discontinuing study treatment. The definition of effective contraception should be in agreement with local regulation and based on the judgment of the principal investigator or a designated associate.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | three to six months
  Time from treatment to death of patients

SECONDARY OUTCOMES:
Side effects of salvage chemotherapy | three to six months
  Side effects of salvage chemotherapy are coded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Quality of life before and after treatment | three to six months
  Quality of life is assessed with EORTC QLQ-C30 (version 3) questionnaire.
body weight in kilograms | three to six months
  body weight in kilograms
body mass index (BMI) in kg/m^2 | three to six months
  body mass index (BMI) in kg/m^2
serum sugar in mg/dL | three to six months
  serum sugar in mg/dL
serum albumin in g/dL | three to six months
  serum albumin in g/dL
serum prealbumin in mg/dL | three to six months
  serum prealbumin in mg/dL
serum total protein in g/dL | three to six months
  serum total protein in g/dL
serum transferrin saturation in % | three to six months
  serum transferrin saturation in %
serum total cholesterol (TC) in mg/mL | three to six months
  serum total cholesterol (TC) in mg/mL
serum low-density lipoprotein cholesterol (LDL-C) in mg/mL | three to six months
  serum low-density lipoprotein cholesterol (LDL-C) in mg/mL
serum high-density lipoprotein cholesterol (HDL-C) in mg/mL | three to six months
  serum high-density lipoprotein cholesterol (HDL-C) in mg/mL
serum triglyceride (TG) in mg/dL | three to six months
  serum triglyceride (TG) in mg/dL
nitrogen balance in grams | three to six months
  nitrogen balance in grams
Performance status | three to six months
  Performance status is documented by Eastern Cooperative Oncology Group (ECOG) scale.
Interleukin 6 (IL-6) in pg/mL | three to six months
  Interleukin 6 (IL-6) in pg/mL
Interleukin 10 (IL-10) in pg/mL | three to six months
  Interleukin 10 (IL-10) in pg/mL
tumor necrosis factor-α (TNF-α) in pg/mL | three to six months
  tumor necrosis factor-α (TNF-α) in pg/mL
C-reactive protein (CRP) in mg/dL | three to six months
  C-reactive protein (CRP) in mg/dL
procalcitonin (PCT) in ng/mL | three to six months
  procalcitonin (PCT) in ng/mL
blood Na in mEq/L | three to six months
  blood Na in mEq/L
blood K in mEq/L | three to six months
  blood K in mEq/L
blood Ca in mg/dL | three to six months
  blood Ca in mg/dL
blood Cl in mEq/L | three to six months
  blood Cl in mEq/L
blood P in mg/dL | three to six months
  blood P in mg/dL
blood aspartate aminotransferase (AST) in U/L | three to six months
  blood aspartate aminotransferase (AST) in U/L
blood alanine aminotransferase (ALT) in U/L | three to six months
  blood alanine aminotransferase (ALT) in U/L
blood gamma-glutamyl transpeptidase (γGT) in U/L | three to six months
  blood gamma-glutamyl transpeptidase (γGT) in U/L
blood direct bilirubin in mg/dL | three to six months
  blood direct bilirubin in mg/dL
blood albumin in g/dL | three to six months
  blood albumin in g/dL
international normalized ratio (INR) | three to six months
  international normalized ratio (INR)
partial thromboplastin time (PTT) in seconds | three to six months
  partial thromboplastin time (PTT) in seconds
leukocyte-count in cells/μL | three to six months
  leukocyte-count in cells/μL
platelet-count in cells/μL | three to six months
  platelet-count in cells/μL
erythrocyte-count in cells/μL | three to six months
  erythrocyte-count in cells/μL
Complications of HPN | three to six months
  Complications of HPN include adverse events (AEs) and severe adverse events (SAEs). AEs and SAEs are coded using the MedDRA system (version 18.0, http://www.meddra.org) and summarized descriptively by system organ class.
Cycles of salvage chemotherapy completed | three to six months
  How many cycles of salvage chemotherapy for unresectable metastatic or recurrent gastric cancer is completed after intervention of HPN

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Yuan Jaw-Yuan, PhD, Study Chair — Kaohsiung Medical University
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No